CLINICAL TRIAL: NCT05806853
Title: Phase II Prospective Monocentric Study on Prostate Cancer Restaging by Using PET/MR With Innovative Radiotracers
Brief Title: PET/MR for Prostate Cancer Restaging: a Phase II Prospective Monocentric Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Maria Picchio, Associate professor, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PCa Restaging- PET/MR
Record Dates: First submitted 2023-03-22; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; biochemical recurrence; PET/MR
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; BAY 86-7548

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dual tracer PET/MRI (Experimental): All patients undergo PET/MRI with 68Ga-PSMA and 68Ga-DOTA-RM2. 68Ga-PSMA dose: 160 +-50 MBq, route of administration: intravenous 68Ga-DOTA-RM2 dose: 140 +-50 MBq, route of administration: intravenous
  Interventions: Drug: 68Ga-PSMA; Drug: 68Ga-RM2

INTERVENTIONS:
Drug: 68Ga-PSMA — Glu-NH-CO-NH-Lys-(Ahx)-[68Ga(HBED-CC)] (68Ga-PSMA)
Drug: 68Ga-RM2 — Bombesin receptor antagonist (68Ga-RM2)

SUMMARY:
The overall goal is to provide an innovative approach to restage patients with biochemical recurrence of prostate cancer by using hybrid PET/MR with innovative radiotracers (68Ga-PSMA and 68Ga-RM2)

DETAILED DESCRIPTION:
Sixty consecutive patients with biochemical recurrence (PSA≥0.2 ng/ml), previously treated with radical prostatectomy for organ confined prostate cancer will be enrolled; patients with previous and/or concomitant androgen deprivation therapy will be excluded from enrolment.

All patients will undergo both 68Ga-PSMA PET/MR and 68Ga-RM2 PET/MR imaging at San Raffaele Scientific Institute in two different days; all clinical and pathological variables available at the time of PET/MR studies will be recorded for each patient.

PET/MR results will be compared to other imaging procedures performed and available in the course of routinely work-up evaluation. Treatment approach will be based on all available clinical and instrumental data, including 68Ga-PSMA and 68Ga-RM2 PET/MR, evaluated during multidisciplinary sessions including expert Urologists, Nuclear Medicine and Radiologist physicians. Patients with local recurrence will be candidate to salvage radiation therapy (sRT). Patients presenting only LN recurrence will be proposed to be submitted to salvage lymph node (LN) dissection (sLND) or sRT; alternatively, conventional androgen deprivation therapy will be performed in those patients who will not be willing to undergo secondary surgery or radiation therapy.

To assess the diagnostic accuracy of 68Ga-PSMA and 68Ga-RM2 PET/MR, images will be validated with: 1) histology (when deemed necessary by the clinician as expected under the normal care pathway) obtained by echographically-guided biopsy in suspected local recurrence or during sLND in the event of suspected nodal recurrence; 2) biochemical response after tailored treatment in patients submitted to sRT for local or LN recurrence 3) conventional imaging modalities performed to assess disease status as part of the routine clinical work-up. 68Ga-PSMA and 68Ga-RM2 PET/MR will be correlated with available clinical and pathological features. To assess the impact of 68Ga-PSMA PET/MR and 68Ga-RM2 PET/MR in changing patients' management, patients will be followed-up after the execution of PET/MR studies. Patients will be followed-up until the end of the study period

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological proven diagnosis of prostate cancer.
* Patients treated with radical therapy (RP o EBRT, with or without further adjuvant therapies), who present rising serum PSA values ≥ 0.2 ng/mL.
* Age ≥ 18 years-old.
* Willing to provide a signed informed consent.

Exclusion Criteria:

* Age < 18 years-old.
* Previous and/or concomitant androgen deprivation therapy will be excluded.
* Any additional medical condition that may significantly interfere with study compliance.
* Contraindications to MR study (i.e. Pacemaker

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the diagnostic accuracy of 68Ga-PSMA PET/MR to identify the site of recurrence in patients with biochemical relapse of PCa after primary treatment and comparison with the performances of 68Ga-RM2 PET/MR | Imaging will be performed at T0 and T1 (at least 2 days apart). PET/MR results will be compared to other imaging procedures performed in the course of routinely work-up evaluation.
  Diagnostic accuracy will be measured by sensitivity, specificity, positive predicted value and negative predicted value

SECONDARY OUTCOMES:
To correlate 68Ga-PSMA PET/MR and 68Ga-RM2 PET/MR imaging with clinical and pathological features. | Imaging will be performed at T0 and T1 (at least 2 days apart). Analysis after enrollment completion
  Univariate and multivariate logistic regression will be used to study the association (measured with odds ratio) between clinical/histopathological data and imaging findings. The clinical/histoapthological data that will be considered are ISUP grade, age (years), time between radical treatment and biochemical recurrence (months), PSA at time of imaging (ng/ml), initial PSA (ng/ml), PSA doubling time and PSA velocity.
To evaluate the results of a lesion-targeted approach in terms of biochemical-recurrence-free survival and clinical recurrence-free survival | 0-36 months
  To assess the impact of 68Ga-PSMA PET/MR and 68Ga-RM2 PET/MR in changing patients' management, patients will be followed-up after the execution of PET/MR studies. Patients will be followed-up until the end of the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/53/NCT05806853/Prot_SAP_000.pdf